CLINICAL TRIAL: NCT01467076
Title: Pilot Randomized Clinical Trial of Inhaled PGE1 in Neonates With Sub-Optimal Response to Inhaled Nitric Oxide
Brief Title: Inhaled Prostaglandin E1 (IPGE1) for Hypoxemic Respiratory Failure (NHRF)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was halted due to futility concerns based on the unmet benchmarks as specified in the pilot study protocol.
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NICHD-NRN-0046; U10HD040689 (NIH); U10HD021385 (NIH); U10HD027904 (NIH); U10HD027880 (NIH); U10HD034216 (NIH); U10HD040492 (NIH); U10HD053109 (NIH); U10HD040461 (NIH); U10HD068263 (NIH); U10HD068270 (NIH); U10HD068278 (NIH); U10HD036790 (NIH)
Record Dates: First submitted 2011-10-17; First posted 2011-11-08 (Estimated); Results first posted 2016-12-30 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Prematurity; Respiratory Insufficiency; Pulmonary Hypertension; Respiratory Distress Syndrome, Newborn
MeSH Terms: conditions — Premature Birth; Respiratory Insufficiency; Hypertension, Pulmonary; Respiratory Distress Syndrome, Newborn | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Inhaled PGE1 (150 ng/kg/min) (Active Comparator): 150 ng/kg/min Inhaled PGE1
  Interventions: Drug: Inhaled PGE1
- Aerosolized Normal Saline (Placebo Comparator): Eligible infants will be randomly assigned to either IPGE1 [150ng/kg/min], IPGE1 [300ng/kg/min] or control group. Infants in the control group will receive the same volume of aerosolized saline and oxygen from the respirator.
  Interventions: Drug: Aerosolized Normal Saline
- Inhaled PGE1 (300 ng/kg/min) (Active Comparator): 300 ng/kg/min of Inhaled PGE1
  Interventions: Drug: Inhaled PGE1

INTERVENTIONS:
Drug: Aerosolized Normal Saline — Two initial doses of IPGE1 will be tested - 150 and 300 ng/kg/min. Thus, there will be three arms to the study - IPGE1 [150], IPGE1 [300], and placebo (normal saline). This design will allow comparison of the two doses of IPGE1 with each other and controls; and also allow comparison of any IPGE1 with controls. Placebo will be administered over a maximum duration of 72 hours.
  Other Names: Normal Saline
  Arms: Aerosolized Normal Saline
Drug: Inhaled PGE1 — Two initial doses of IPGE1 will be tested - 150 and 300 ng/kg/min. Thus, there will be three arms to the study - IPGE1 [150], IPGE1 [300], and placebo (normal saline). This design will allow comparison of the two doses of IPGE1 with each other and controls; and also allow comparison of any IPGE1 with controls. In this Pilot RCT, two doses of IPGE1 (300 and 150 ng/kg/min) will be administered over a maximum duration of 72 hours to determine the optimal dose and duration of therapy.
  Other Names: Inhaled Prostaglandin E1
  Arms: Inhaled PGE1 (150 ng/kg/min); Inhaled PGE1 (300 ng/kg/min)

SUMMARY:
This is a randomized controlled trial (RCT) on the use of Inhaled prostaglandin E1 (IPGE1) in Neonatal Hypoxemic Respiratory Failure (NHRF). Fifty patients recruited at 10 high volume sites within the NICHD Neonatal Research Network will constitute a pilot sample to evaluate the feasibility and safety of prolonged IPGE1 administration and determination of optimal dose. In this Pilot RCT, two doses of IPGE1 (300 and 150 ng/kg/min) will be administered over a maximum duration of 72 hours and compared with placebo. Once feasibility and safety of IPGE1 administered over 72 hours has been demonstrated in the pilot trial, a full scale randomized controlled trial will be planned.

DETAILED DESCRIPTION:
Hypoxemic respiratory failure in the newborn (NHRF) is usually associated with widespread vasoconstriction of the pulmonary microvasculature giving rise to intra- and extra-pulmonary shunts and profound hypoxemia. The goal of therapy is to decrease the regional pulmonary vascular resistance of ventilated lung areas thus decreasing intrapulmonary shunting and selectively reducing the pulmonary-artery pressure without causing systemic vasodilation. Intravenously administered vasodilators lack pulmonary selectivity leading to systemic side effects. Inhaled nitric oxide (INO), a selective pulmonary vasodilator, has revolutionized the treatment of respiratory failure in the newborn. However, there is lack of sustained improvement in 30-46% of infants; moreover, INO requires specialized systems for administration, making the treatment expensive. Aerosolized prostaglandins I2 and E1 have been reported to be effective selective pulmonary vasodilators in animals and human adults. In addition, inhaled prostaglandin I2 (IPGI2) has also been reported to be effective in preterm and term newborns, and children with pulmonary hypertension. Although intravenous PGE1 is widely used in neonates, the use of the inhaled form has not been reported in newborns with pulmonary hypertension. Compared to PGI2, PGE1 has a shorter half-life, lower acidity constant (pKa) (6.3 versus 10.5), bronchodilator action, anti-proliferative and anti-inflammatory effects on the alveolar, interstitial and vascular spaces of the lung. Prostaglandin nebulization can be used without the sophisticated technical equipment needed for controlled NO inhalation and hence is less expensive. It has no known toxic metabolites or toxic effects. Prostaglandins and nitric oxide (NO) relax the vascular smooth muscles through two different second-messenger systems; therefore, in combination, INO and IPGE1 may have synergistic effect. The existing literature suggests that inhaled PGE1 is a potential effective vasodilator in the treatment of NHRF . We have reported the safety and feasibility of short-term administration of inhaled PGE1 in an un-blinded Phase I/II dose-escalation study. Four doses ranging from 25 to 300 ng/kg/min were tested for a maximum duration of 3 hours. We have also reported the stability of IPGE1, its emitted dose and aerosol particle size distribution (APSD) in a neonatal ventilator circuit. In addition we have demonstrated the safety of high dose IPGE1 (1200 ng/kg/min) over 24 hours in ventilated piglets. In the current protocol, we propose a pilot to evaluate the feasibility and safety of prolonged IPGE1 in NHRF. Two doses of IPGE1 (300 and 150 ng/kg/min) will be tested followed by weaning for a maximum duration of 72 hours to determine feasibility, safety, optimal dose and duration of therapy in 50 patients in ten NICHD NRN sites. An IND status has been approved by the FDA for this trial.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age less than or equal to 34 weeks
* Postnatal age less than or equal to 7 days (168 hours).
* Assisted ventilation for hypoxemic respiratory failure.
* Diagnosis of NHRF including perinatal aspiration syndrome (meconium, blood, or amniotic fluid), suspected/proven pneumonia/sepsis, respiratory distress syndrome, idiopathic persistent pulmonary hypertension of the newborn (PPHN) or suspected pulmonary hypoplasia.
* Receiving INO for at least 1 hour and not >72 hours.
* Oxygenation Index (OI ) ≥ 15 on any 2 arterial blood gases 15 minutes to 12 hours apart while on INO.
* An indwelling arterial line is present

Exclusion Criteria:

* Any infant in whom a decision has been made not to provide full treatment (e.g. chromosomal anomalies, severe birth asphyxia).
* Known structural congenital heart disease except patent ductus arteriosus and atrial/ventricular level shunts.
* Congenital diaphragmatic hernia.
* Thrombocytopenia unresponsive to platelet transfusion.
* Enrollment in a conflicting and/or Investigational New Drug (IND) clinical trial.

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beena Sood, MD, Principal Investigator — Wayne State University; Martin Keszler, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; C. Michael Cotten, MD, Principal Investigator — Duke University; Abhik Das, PhD, Principal Investigator — RTI International; Krisa P Van Meurs, MD, Principal Investigator — Stanford University; Namasivayam Ambalavanan, MD, Principal Investigator — University of Alabama at Birmingham; Jonathan M Klein, MD, Principal Investigator — University of Iowa; Robin Ohls, MD, Principal Investigator — University of New Mexico; Pablo J Sanchez, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Satyan Lakshminrusimha, MD, Principal Investigator — University of Rochester; Uday Devaskar, MD, Principal Investigator — University of California, Los Angeles; Leif Nelin, MD, Principal Investigator — Research Institute at Nationwide Children's Hospital
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California - Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of Iowa, Iowa City, Iowa
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - Duke University, Durham, North Carolina
  - Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

REFERENCES:
- [Derived] Sood BG, Keszler M, Garg M, Klein JM, Ohls R, Ambalavanan N, Cotten CM, Malian M, Sanchez PJ, Lakshminrusimha S, Nelin LD, Van Meurs KP, Bara R, Saha S, Das A, Wallace D, Higgins RD, Shankaran S; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Inhaled PGE1 in neonates with hypoxemic respiratory failure: two pilot feasibility randomized clinical trials. Trials. 2014 Dec 12;15:486. doi: 10.1186/1745-6215-15-486. PMID 25496504
- See also: Neonatal Research Network — https://neonatal.rti.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Opened for recruitment on 10/20/2011. There was a lag of 33 to 90 days between IRB approval and site readiness to enroll patients. 46 infants were screened at 8 sites, 14 met eligibility criteria, and 7 were randomized. Enrollment was halted for lack of feasibility in mid-May 2012; at that time, only 7 patients had been enrolled.
Pre-assignment Details: Seven eligible infants were not enrolled because parents were unavailable or refused consent for 3 of the infants, 3 infants met ECMO criteria, and 1 had cardio-respiratory arrest.
Groups:
- Control: Aerosolized saline
- Low Dose IPGE1: 150 ng/kg/min
- High Dose IPGE1: 300 ng/kg/min
Period: Overall Study
Arm/Group | Control | Low Dose IPGE1 | High Dose IPGE1
Started | 3 | 2 | 2
Completed | 2 | 2 | 2
Not Completed | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Infants randomized to the Control group were given the placebo dose.
  Infants randomized to the Low Dose IPGE1 were given the lower dose.
  Infants randomized to the High Dose IPGE1 were given the higher dose.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Low Dose IPGE1 | High Dose IPGE1 | Total
Number analyzed (Participants) | 3 | 2 | 2 | 7
Age, Customized [Mean (Full Range); unit: hours]
  Age at Randomization | 41.75 [27.80 to 58.33] | 11.30 [7.10 to 15.50] | 26.65 [10.28 to 43.03] | 28.73 [7.10 to 58.33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 4
  Male | 2 | 1 | 0 | 3
Birthweight [Mean (Full Range); unit: grams] | 3591 [2880 to 3965] | 3530 [3470 to 3590] | 3320 [3103 to 3537] | 3496 [2880 to 3965]
Delivery by Cesarean Section [Number; unit: participants] | 2 | 2 | 1 | 5
Intubation in Delivery Room [Number; unit: participants] | 0 | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Feasibility Assessed as the Number of Participants Who Were Enrolled in the Study
Description: The primary outcome is the ability to recruit adequate number of infants (n=50) in a 9 month period without excessive (>20%) protocol violations.
Time Frame: From study start through 9 months after 75% of the participating sites are enrolling
Population: Late preterm & term infants ≤ 7 days postnatal age undergoing conventional ventilation (CNV) or high frequency oscillatory ventilation (HFOV) for NHRF (including perinatal aspiration syndrome, suspected/proven pneumonia/sepsis, respiratory distress syndrome, idiopathic PPHN or suspected pulmonary hypoplasia) with suboptimal response to INO
Measure: Number; unit: participants
Arm/Group | Control | Low Dose IPGE1 | High Dose IPGE1
Number analyzed (Participants) | 3 | 2 | 2
participants | 3 | 2 | 2

2. Secondary Outcome: Change in Partial Pressure of Oxygen in the Blood (PaO2)
Description: Changes in PaO2 based on the arterial blood gases (ABG) measurements obtained after 60 minutes and ABG obtained 4 hours after start of study aerosol.
Time Frame: Measurement of ABG at 60±15 minutes and 4±2 hours after start of study aerosol.
Population: To gauge the improvement in PaO2 for each group, the average of the difference between the two PaO2 ABG measurements (measurement at 4±2 hours-measurement at 60±15 minutes after start of study aerosol) and the range(minimum, maximum) of the differences between OI ABG measurements at the two time points within each group are presented here.
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Control | Low Dose IPGE1 | High Dose IPGE1
Number analyzed (Participants) | 3 | 2 | 2
mmHg | 30 [-1 to 59] | 85 [22 to 148] | 48 [-9 to 95]

3. Secondary Outcome: Change in Oxygenation Index (OI)
Description: Change in OI based on the arterial blood gases (ABG) measurements obtained at 60±15 minutes and ABG obtained 4±2 hours after start of study aerosol.
Time Frame: Measurement of ABG at 60±15 minutes and 4±2 hours after start of study aerosol.
Population: To gauge change in OI for each group we present both the average and the range of the difference between the two OI ABG measurements (measurement at 4±2 hours - measurement at 60±15 minutes after start of study aerosol). A positive difference indicates an increase in OI measurement; a negative difference indicates a decrease in OI measurement.
Measure: Mean (Full Range); unit: oxygenation index
Arm/Group | Control | Low Dose IPGE1 | High Dose IPGE1
Number analyzed (Participants) | 3 | 2 | 2
oxygenation index | 4 [-1 to 9] | 14 [6 to 21] | 10 [-5 to 25]

4. Secondary Outcome: Need for Inhaled Nitric Oxide (INO) 72 Hours After INO
Description: Administration of INO continued after the Infant was on INO for 72 hours
Time Frame: Date of first administration of INO to date of final discontinuation of INO
Population: Date of final discontinuation of INO was not available for 1 infant in the Control group and 1 infant in the LOW DOSE IPGE1 group
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Low Dose IPGE1 | High Dose IPGE1
Number analyzed (Participants) | 2 | 1 | 2
Participants | 1 | 0 | 0

5. Secondary Outcome: Duration of iNO Therapy
Description: Duration the infant is on INO from initial administration of INO to final discontinuation of INO.
Time Frame: From date of first administration of INO to date of final discontinuation of INO.
Population: The date of final discontinuation of INO was recorded for 2 infants in the control group, 1 infant in the low dose and all 2 infants in the high dose group.
Measure: Mean (Full Range); unit: hours
Arm/Group | Control | Low Dose IPGE1 | High Dose IPGE1
Number analyzed (Participants) | 2 | 1 | 2
hours | 59.02 [44.95 to 73.08] | 18.57 [18.57 to 18.57] | 56.22 [50.35 to 62.08]

6. Secondary Outcome: Death
Description: Deaths prior to discharge home.
Time Frame: From birth through status (death, transfer, or discharge).
Population: All 3 infants in the control group, 2 infant in the Low dose and 2 infants in the High dose IPGE1 groups have status data (death, transfer or discharge).
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Low Dose IPGE1 | High Dose IPGE1
Number analyzed (Participants) | 3 | 2 | 2
Participants | 0 | 0 | 0

7. Secondary Outcome: Need for Extracorporeal Membrane Oxygenation (ECMO)
Description: ECMO provided at the institution for the infant after discontinuation of study aerosol.
Time Frame: From after discontinuation of study aerosol through status (death, transfer, or discharge).
Population: All 3 infants in the control group, 2 infant in the Low dose and 2 infants in the High dose IPGE1 groups have data on ECMO use at the institution after discontinuation of study aerosol.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Low Dose IPGE1 | High Dose IPGE1
Number analyzed (Participants) | 3 | 2 | 2
Participants | 2 | 1 | 2

8. Secondary Outcome: Duration of Mechanical Ventilation
Description: Duration the infant is on Mechanical Ventilation from birth through status (death, transfer or discharge)
Time Frame: From birth through status (death, transfer or discharge)
Population: All 3 infants in the aerosolized saline group, and the 2 infants in the lower dose IPGE1 group and high dose IPGE1 Group have the number of days on mechanical ventilation from birth to death, transfer or discharge.
Measure: Mean (Full Range); unit: Days
Arm/Group | Control | Low Dose IPGE1 | High Dose IPGE1
Number analyzed (Participants) | 3 | 2 | 2
Days | 22 [17 to 30] | 8 [4 to 11] | 16 [13 to 19]

9. Secondary Outcome: Number of Days of Supplemental Oxygen (O2) Used
Description: Number of days from birth during which the FiO2 at some point was > 0.21.
Time Frame: From birth through status (death, transfer or discharge)
Population: All 3 infants in the aerosolized saline group, and the 2 infants in the lower dose IPGE1 group and high dose IPGE1 Group have the number of days on supplemental oxygen from birth to death, transfer or discharge.
Measure: Mean (Full Range); unit: Days
Arm/Group | Control | Low Dose IPGE1 | High Dose IPGE1
Number analyzed (Participants) | 3 | 2 | 2
Days | 43 [24 to 79] | 8 [4 to 12] | 11 [9 to 13]

10. Secondary Outcome: Length of Hospital Stay
Description: Length of stay in hospital from birth to discharge home.
Time Frame: From birth to discharge home
Population: Two infants in the aerosolized saline group, and 2 infants in the lowd ose IPGE1 group and high dose IPGE1 Group were discharged home/chronic care.
Measure: Mean (Full Range); unit: Days
Arm/Group | Control | Low Dose IPGE1 | High Dose IPGE1
Number analyzed (Participants) | 3 | 2 | 2
Days | 64 [27 to 81] | 31 [21 to 40] | 39 [29 to 49]

ADVERSE EVENTS:
Time Frame: Enrolled infants were monitored continuously throughout study aerosol administration and through 48 hours post study aerosol discontinuation for possible adverse effects of PGE1.
Description: Monitored adverse events (AEs) include arrhythmia, hypotension, seizures, bleeding tendency, diarrhea, and seizures.
Arm/Group | Control | Low Dose IPGE1 | High Dose IPGE1
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=3) | Low Dose IPGE1 (N=2) | High Dose IPGE1 (N=2)
Hypotension (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — One infant in the control group developed moderate hypotension 66 hours after initiation of the study aerosol. It was completely resolved within an hour of its onset. The even was not attributed to study aerosol.
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0)
New onset seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0)
New onset bleeding (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0)
Fever (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) — One infant in the control group developed transient, self-resolved mild fever within 5 minutes of starting the study aerosol which was completely resolved within 6 hours after onset. The event was not attributed to study aerosol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators must adhere to the Neonatal Research Network Publication policies.